CLINICAL TRIAL: NCT06938230
Title: Promoting A School Culture of Safety in the Era of COVID-19: Assessing Feasibility and Impact of a Health Education Initiative
Brief Title: Coronavirus Disease of 2019 (COVID-19) Health Education Initiative for School Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lisa Gwynn, Full Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20220254; 1OT2HD108111-01 (NIH)
Record Dates: First submitted 2025-04-17; First posted 2025-04-22 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education Initiative (Experimental): Participants will receive the health education session for up to 6 months.
  Interventions: Behavioral: Health Education Initiative
- Control Group (No Intervention): Participants in this group will not receive any health education and total participation is up to 6 months.

INTERVENTIONS:
Behavioral: Health Education Initiative — Participants will receive a one time 45 minute intervention session. During the session participants will receive information regarding COVID-19 disease process and behavioral effects and had the opportunity to ask questions.
  Arms: Health Education Initiative

SUMMARY:
The purpose of this study is to compare COVID-19 knowledge, experiences, and health behaviors between participants who received the health initiative and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of students enrolled in:
* Arch Creek Elementary, Fulford Elementary
* Greynolds Park Elementary
* Sabal Palm Elementary
* North Miami Middle school,
* John F Kennedy (JFK) Middle School
* North Miami Senior High
* North Miami Beach High
* Booker T. Washington High
* Able to read and write in English, Spanish, or Creole at a 5th grade level

Exclusion criteria:

* Does not speak:
* English
* Spanish
* Creole

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Gwynn, DO, Principal Investigator — University of Miami; Elizabeth Pulgaron, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Education Initiative | Control Group
Started | 76 | 36
Completed | 20 | 18
Not Completed | 56 | 18
Not completed — Lost to Follow-up | 56 | 18

BASELINE CHARACTERISTICS:
Population: Baseline measures including age, sex, ethnicity and race were optional for participants to report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Education Initiative | Control Group | Total
Number analyzed (Participants) | 76 | 36 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There were only 64 participants analyzed because the remaining participants did not respond to the question.
  years
    number analyzed (Participants) | 29 | 35 | 64
    (all) | 44.34 (8.80) | 41.69 (7.85) | 42.89 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were only 65 participants analyzed, because the remaining participants did not respond to the question.
  Participants
    number analyzed (Participants) | 29 | 36 | 65
    Female | 26 | 32 | 58
    Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 17 | 31 | 48
  Unknown or Not Reported | 52 | 0 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 28 | 46
  White | 8 | 5 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 49 | 2 | 51

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Acceptability of Intervention as Measured by Acceptability Questionnaire
Description: Scores range from 1 ("strongly disagree") to 5 ("strongly agree"), with higher scores indicating more knowledge, value, application, or satisfaction. Evaluation was collected directly after the intervention, at baseline.
Time Frame: Baseline
Population: This was data collection only for the health education initiative. The control group did not participate in this section.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Initiative
Number analyzed (Participants) | 76
score on a scale | 4.47 (0.89)

2. Primary Outcome: Evaluation of Confidence in COVID Healthcare Decision Making as Measured by COVID Confidence Questionnaire
Description: Scores range from 1 ("strongly disagree") to 5 ("strongly agree"), with higher scores indicating more knowledge, value, application, or satisfaction.
Time Frame: 6 months
Population: This was only administered to the intervention group. No control participants were analyzed because they did not receive this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Initiative
Number analyzed (Participants) | 76
score on a scale | 4.38 (0.86)

3. Primary Outcome: Number of Caregivers Who Received COVID-19 Vaccine
Description: The unit of measure is the number of caregivers who received COVID-19 vaccine at baseline
Time Frame: Baseline
Population: The number of participants analyzed at 6 months is lower than those who were analyzed at baseline due to participants lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 49 | 34
Participants | 35 | 24

4. Primary Outcome: Number of Children Who Received COVID-19 Vaccine
Description: unit of measure number of children
Time Frame: Baseline
Population: The number of participants analyzed at baseline differs from the number analyzed at 6 months because participants were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 52 | 35
Participants | 23 | 18

5. Primary Outcome: Health Behaviors as Measured by Health Behavior Questionnaire
Description: Scores range from 1 ("strongly disagree") to 5 ("strongly agree"), with higher scores indicating greater intent to engage in health behaviors to prevent COVID-19.
Time Frame: Baseline
Population: The number of participants analyzed differ between baseline and 6 months because participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 61 | 34
score on a scale | 4.10 (1.10) | 3.76 (1.37)

6. Primary Outcome: Number of Caregivers Who Received COVID-19 Vaccine
Description: The unit of measure is the number of caregivers who received COVID-19 vaccine
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 29 | 17
Participants | 18 | 7

7. Primary Outcome: Health Behaviors as Measured by Health Behavior Questionnaire
Description: as for outcome 5
Time Frame: 6 month
Population: The number of participants analyzed differ between baseline and 6 months because participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 33 | 18
score on a scale | 4.09 (0.82) | 3.96 (1.18)

8. Secondary Outcome: PTSD as Measured by the University of California Los Angeles (UCLA) Brief COVID-19 Screen for Child/Adolescent Post Traumatic Stress Disorder (PTSD)
Description: Individual item scores range from 0 to 4, individual total sum scores range from 0 to 44 higher scores indicate more symptoms of PTSD. Total sum score ranging from 1-10 is considered "minimal PTSD", total sum score ranging from 11-20 is considered "mild PTSD", total sum scores of 21 or more is considered "potential PTSD".
Time Frame: Baseline, 6 month follow up
Population: The number of participants analyzed at baseline is lower than the overall number of participants, because some participants did not complete their packet of questionnaires, including the present measure. There were fewer participants at the 6-month follow-up because participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 29 | 35
score on a scale
  Baseline | 5.83 (6.49) | 5.77 (8.63)
  6 month follow up: number analyzed (Participants) | 18 | 19
  6 month follow up | 4.6 (6.7) | 7.74 (8.27)

9. Secondary Outcome: COVID Anxiety as Measured by the Coronavirus Anxiety Scale
Description: individual item score ranges from 0 to 4, individual total sum scores range from 0 to 20 higher scores indicate more symptoms of COVID specific anxiety. Total sum scores of greater than of equal to 9 equals "probable dysfunctional Coronavirus related anxiety".
Time Frame: Baseline, 6 month follow up
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 29 | 35
score on a scale
  Baseline | 0.21 (0.62) | 1.37 (3.95)
  6 month follow up: number analyzed (Participants) | 18 | 19
  6 month follow up | 0.83 (2.28) | 0.42 (1.22)

10. Primary Outcome: Number of Children Who Received COVID-19 Vaccine
Description: unit of measure number of children
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education Initiative | Control Group
Number analyzed (Participants) | 28 | 16
Participants | 11 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Health Education Initiative | Control Group
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/36
Other Adverse Events (participants affected / at risk) | 0/76 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT06938230/Prot_000.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT06938230/ICF_001.pdf